CLINICAL TRIAL: NCT02147171
Title: The Bioavailability of Retinal Carotenoids in the Older Human Eye and Their Effects on Photoreceptor Performance
Brief Title: Carotenoid Supplementation and Normal Ocular Health
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Manchester (Other)
Responsible Party: Principal Investigator, Laura Patryas, Miss, University of Manchester
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: BB/F017227/1
Record Dates: First submitted 2014-04-16; First posted 2014-05-26 (Estimated); Last update posted 2014-05-26 (Estimated); Status verified 2014-04

CONDITIONS: Retinal Ageing
Keywords: Retinal ageing, macular pigment, visual function

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Active lutein group (Active Comparator): 44 participants taking VisionAce daily for a period of 1 year
  Interventions: Dietary Supplement: VisionAce
- Placebo group (Placebo Comparator): 44 participants taking placebo daily for a period of 1 year
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: VisionAce
  Arms: Active lutein group
Dietary Supplement: Placebo
  Arms: Placebo group

SUMMARY:
Normal ageing affects vision as a result of preretinal and retinal changes. Photoreceptors, the light sensitive cells in the retina, degenerate and the rods (responsible for night vision) are most susceptible to damage with increasing age. Rod loss leads to poor vision in the dark which increases the risk of accidents amongst the elderly. Macular pigment (located in the photoreceptors)is thought to protect the retina and reduce the risk of age related changes. Dark adaptation, mediated by the rods, slows down with age, and is also reduced in AMD (age-related macular degeneration). Recent evidence suggests that lutein (the main component of macular pigment) supplementation improves the dark adaptation deficit in AMD subjects. Research into the effects of lutein in a normal human has not been previously conducted. Since the older population is increasing, our aim is to firstly establish the extent of night vision loss (using dark adaptometry) and secondly to examine the possibility of slowing down or reversing this loss through lutein supplementation.

DETAILED DESCRIPTION:
It is believed that the macular pigment protects the retina against photooxidative damage which can lead to agerelated macular degeneration (AMD). It is also hypothesized to enhance visual performance in normal human eyes. Much of the research into lutein supplementation has been centered around AMD subjects. AMD can result from agerelated retinal photoreceptor dysfunction which could hypothetically be prevented or slowed down through early supplementation. To our knowledge, the effects of lutein in normal ageing, have not been studied previously.

Macular pigment is composed of lutein and zeaxanthin. These compounds absorb blue light and therefore protect the retinal photoreceptors. They also possess powerful antioxidant properties and therefore help maintain the integrity of the macular region. With increasing age, the visual performance worsens as a result of preretinal and retinal changes such as photoreceptor degeneration. Rods (responsible for night vision) are highly susceptible to degeneration in a normal aging eye and in AMD. Older subjects often complain of reduced vision in the dark which can contribute to increased risk of road traffic accidents and falls. Since the older population is rapidly growing, it is vital to study the mechanics of photoreceptor degeneration and the possible beneficial effects of supplementation with retinal carotenoids, particularly lutein.

The supplement that will be used in this study will be the commercially available Visionace Plus (details attached). The manufacturer of Visionace Plus is Vitabiotics. The placebo will be soya-based, also manufactured by Vitabiotics.

ELIGIBILITY:
Inclusion Criteria:

1. Not on food supplements containing lutein or zeaxanthin
2. Visual acuity at least 0.4 logMAR units (6/15 Snellen)

4. Body mass index of less than 35 5. No diagnosed ocular disease (e.g. established AMD, cataract, glaucoma) 6. Age between 50 and 90

Exclusion Criteria:

1. Diabetes
2. Any diagnosed ocular disease (e.g. AMD, cataract, glaucoma)
3. Under 50 and over 90 years old

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2011-11; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Changes in macular pigment optical density | 12 months
Changes in serum lutein | 12 months

SECONDARY OUTCOMES:
Changes in visual performance | 12 months
  The following parameters of visual function will be assessed:
  Visual acuity Contrast Sensitivity Resolution limit Dark adaptation

CONTACTS AND LOCATIONS:
Overall Officials: Ian Murray, Study Director — University of Manchester
Locations (1):
- University of Manchester, Manchester, United Kingdom